CLINICAL TRIAL: NCT01744964
Title: Alterations in the Ability to Tolerate Experimental Pain by Apomorphine and Its Association With a Dopamine Transporter Polymorphism
Brief Title: Apomorphine Effects on Experimental Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 0078-09-RBM
Record Dates: First submitted 2012-12-06; First posted 2012-12-07 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: apomorphine; dopamine transporter gene; SLC6A3; cold pressor test; tolerance; experimental pain; dopamine agonist
MeSH Terms: interventions — Apomorphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator): Assessment of experimental pain models before and after treatment
  Interventions: Drug: Apomorphine
- Apomorphine (Active Comparator): Assessment of experimental pain models before and after treatment
  Interventions: Drug: Apomorphine

INTERVENTIONS:
Drug: Apomorphine — 1.5 mg Apomorphine
  Other Names: Active Comparator: Apomorphine

SUMMARY:
The aims of this study were to assess the effects of the dopamine agonist apomorphine on experimental pain models in healthy subjects and to explore the possible association between these effects and a common polymorphism within the dopamine transporter gene.

DETAILED DESCRIPTION:
Healthy volunteers (n=105) participated in this randomized double-blind, placebo-controlled, cross-over trial. Heat pain threshold and intensity, cold pain threshold, and the response to tonic cold pain (latency, intensity, and tolerance) were evaluated before and for up to 120 min after the administration of 1.5 mg apomorphine/placebo. A polymorphism (DAT-1) within the dopamine transporter gene (SLC6A3) was investigated.

ELIGIBILITY:
Inclusion Criteria:

- healthy and free from chronic pain of any type did not use any medications other than oral contraceptives were able to understand the purpose and instructions of the study.

Exclusion Criteria:

- any type of medical or painful condition use of medications or recreational drugs pregnancy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Cold pain tolerance | 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Elon Eisenberg, MD, Principal Investigator — Rambam Health Care Campus, Haifa, Israel
Locations (1):
- Rambam Health Care Campus, Haifa, Israel